CLINICAL TRIAL: NCT03962244
Title: Endoscopic Management of ESOphago-gastric Anastomotic LEAKages (EsoLeak): Stent Therapy Versus Endoscopic Vacuum Therapy
Brief Title: Stent Therapy Versus Endoscopic Vacuum Therapy for Anastomotic Leaks After Esophagectomy
Acronym: EsoLeak
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital of Cologne (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Seung-Hun Chon, PI, University Hospital of Cologne
Other Study IDs: 19-1201
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Leaks, Anastomotic
Keywords: Esophagectomy, Esophageal Cancer, Vacuum therapy, Stents
MeSH Terms: conditions — Anastomotic Leak; Esophageal Neoplasms | interventions — Negative-Pressure Wound Therapy; Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SEMS Group: The outcome of using self-expanding metal stents (SEMS) in the treatment of postoperative leakage after esophagogastrostomy
  Interventions: Device: Self-Expanding Metal Stent
- EVT Group: The outcome of using endoscopic vacuum therapy (EVT) in the treatment of postoperative leakage after esophagogastrostomy
  Interventions: Device: EsoSponge

INTERVENTIONS:
Device: EsoSponge — Endoscopically placed an EsoSponge for Negative pressure wound therapy in the area of the esophagogastric anastomotic leaks
  Other Names: Negative pressure wound therapy
  Groups: EVT Group
Device: Self-Expanding Metal Stent — Endoscopically placed self-expanding-metal-stent (SEMS) for negative pressure wound therapy in the area of the esophagogastric anastomotic leaks
  Other Names: SEMS, stent
  Groups: SEMS Group

SUMMARY:
Exploratory study of the efficiency of endoscopic stenting versus endoscopic vacuum therapy in patients with intrathoracic esophago-gastric anastomotic leakage after oncological resection of the esophagus.

DETAILED DESCRIPTION:
We analyze the outcome of using self-expanding metal stents (SEMS) and endoscopic vacuum therapy (EVT) in the treatment of postoperative leakage after esophagogastrostomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed oesophageal carcinoma or similarly operated neoplasia (e.g., GIST, NET, subepithelial tumors)
* Esophagectomy with an intrathoracic esophago-gastric anastomosis
* Radiologically or endoscopically diagnosed esophago-gastric anastomotic leakage
* Clinical symptoms / symptoms due to insufficiency or increase in signs of inflammation, most likely as a result of anastomotic leakage
* Age ≥18 years
* To empower the patient to understand the scope of the study and its consequences or information, to consent to it and to sign the educational documents.
* Written declaration of consent of the patient to be included. If the patient is unable to sign by hand, a witness must confirm the oral examination by signature.

Exclusion Criteria:

* Macroscopically incompletely resected tumor (R2), palliative resection
* Endoscopically verified necrosis or critical ischemia of the anastomotic region of the interponate
* Size of insufficiency more than 50% of circumference
* Impossibility of radiological interventional insertion of a drainage
* Early anastomotic leak (≤ 48 hours postoperatively), late insufficiencies (> 4 weeks)
* Therapeutic anticoagulation
* Severe septic shock that indicates surgical therapy
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an intrathoracic esophago-gastric anastomotic leak after oncologic esophagectomy (Ivor-Lewis).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction of treatment assessed by EORTC QLQ - OES18 | 6 months
  Assessing the quality of life of patients during the treatment of stent and EVT with a questionnaire by EORTC QLQ - OES18. This Questionnaire was developed to assess the quality of life of cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hun Chon, MD, Principal Investigator — University Hospital of Cologne; Michael Tachezy, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf (UKE)
Locations (2):
- Germany (2):
  - University Hospital of Cologne, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bartella I, Mallmann C, Burger M, Toex U, Goeser T, Bruns C, Chon SH. Stent-over-sponge (SOS): a rescue option in patients with complex postoperative anastomotic leaks after esophagectomy. Endoscopy. 2019 Aug;51(8):E227-E228. doi: 10.1055/a-0885-9659. Epub 2019 May 2. No abstract available. PMID 31049889
- [Result] Berlth F, Bludau M, Plum PS, Herbold T, Christ H, Alakus H, Kleinert R, Bruns CJ, Holscher AH, Chon SH. Self-Expanding Metal Stents Versus Endoscopic Vacuum Therapy in Anastomotic Leak Treatment After Oncologic Gastroesophageal Surgery. J Gastrointest Surg. 2019 Jan;23(1):67-75. doi: 10.1007/s11605-018-4000-x. Epub 2018 Oct 29. PMID 30374816
- [Result] Grimminger PP, Goense L, Gockel I, Bergeat D, Bertheuil N, Chandramohan SM, Chen KN, Chon SH, Denis C, Goh KL, Gronnier C, Liu JF, Meunier B, Nafteux P, Pirchi ED, Schiesser M, Thieme R, Wu A, Wu PC, Buttar N, Chang AC. Diagnosis, assessment, and management of surgical complications following esophagectomy. Ann N Y Acad Sci. 2018 Dec;1434(1):254-273. doi: 10.1111/nyas.13920. Epub 2018 Jul 8. PMID 29984413
- [Result] Chon SH, Toex U, Plum PS, Fuchs C, Kleinert R, Bruns C, Goeser T. Successful closure of a gastropulmonary fistula after esophagectomy using the Apollo Overstitch and endoscopic vacuum therapy. Endoscopy. 2018 Jul;50(7):E149-E150. doi: 10.1055/a-0592-6384. Epub 2018 Apr 13. No abstract available. PMID 29653446
- [Result] Bludau M, Fuchs HF, Herbold T, Maus MKH, Alakus H, Popp F, Leers JM, Bruns CJ, Holscher AH, Schroder W, Chon SH. Results of endoscopic vacuum-assisted closure device for treatment of upper GI leaks. Surg Endosc. 2018 Apr;32(4):1906-1914. doi: 10.1007/s00464-017-5883-4. Epub 2017 Dec 7. PMID 29218673
- [Derived] Mandarino FV, Barchi A, Leone L, Fanti L, Azzolini F, Viale E, Esposito D, Salmeri N, Puccetti F, Barbieri L, Cossu A, Treppiedi E, Elmore U, Rosati R, Danese S. Endoscopic vacuum therapy versus self-expandable metal stent for treatment of anastomotic leaks < 30 mm following oncologic Ivor-Lewis esophagectomy: a matched case-control study. Surg Endosc. 2023 Sep;37(9):7039-7050. doi: 10.1007/s00464-023-10213-8. Epub 2023 Jun 23. PMID 37353654
- [Derived] Tachezy M, Chon SH, Rieck I, Kantowski M, Christ H, Karstens K, Gebauer F, Goeser T, Rosch T, Izbicki JR, Bruns CJ. Endoscopic vacuum therapy versus stent treatment of esophageal anastomotic leaks (ESOLEAK): study protocol for a prospective randomized phase 2 trial. Trials. 2021 Jun 2;22(1):377. doi: 10.1186/s13063-021-05315-4. PMID 34078426